CLINICAL TRIAL: NCT01138241
Title: Incidence and Predictor of TDF Associated Nephrotoxicity and Pharmacokinetic of TDF in HIV-1 Infected Thai Patients: A Sub-study of HIV-NAT 006 Long Term Cohort
Brief Title: Tenofovir Renal Toxicity and Glomerular Filtration Rate (GFR) Validation
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 114
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Renal Function; HIV Infection
Keywords: HIV; Chronic kidney disease; Glomerular Filtration Rate (GFR); Tenofovir; Serum creatinine (sCr); 24 hr urine creatinine clearance; Serum Cystatin C[40]; Modification of Diet in Renal Disease (MDRD); Cockcroft Gault Equation; Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI); 99mTc-diethylenetriaminepentaacetic acid (Tc-99m DTPA) scan; Validate which renal function assessments can accurately detect GFR and assess the effect of TDF concentration on renal function
MeSH Terms: conditions — HIV Infections; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — PBMC collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: ARV experience (TDF based HAART)
  Interventions: Other: Tc99mDTPA renal clearance
- 2: ARV experience (non TDF based ART)
  Interventions: Other: Tc99mDTPA renal clearance
- 3: ARV Naive
  Interventions: Other: Tc99mDTPA renal clearance

INTERVENTIONS:
Other: Tc99mDTPA renal clearance — Tc99mDTPA renal clearance only for 200 patients
  1. Plasma and urine 24 hr for creatinin, glucose, Creatinin clearance, Phosphatemia, uric acid, HCO3, protein, Microalbuminuria, ß2- microglobulinuria
  2. serum creatinine prior and during TDF
  3. TDF plasma levels ( only TDF use) using a validated high-performance liquid chromatography (HPLC)-mass method and stored PBMC for intracellular TDF levels
  4. stored samples (PBMC) for pharmacogenomic study of transporter gene ie Organic Acid Transporter (OAT)
  5. serum for cystanin C ( stored sample prior taking ARV and present time)
  6. intensive 24 hours pharmacokinetic study of TDF in 20 patients

SUMMARY:
To assess and validate equation eGFR in HIV-infected subjects and -uninfected Thai patients

DETAILED DESCRIPTION:
With significant reductions in mortality and risk of progression to AIDS with antiretroviral therapy (ART), complications of long-standing HIV infection and treatment, including renal disease, have become increasingly important. Aging, concomitant metabolic diseases, and use of potentially nephrotoxic ART lead to higher risk for renal disease in HIV-infected persons.WHO encourage TDF as first line ARV regimen. The data on TDF related renal toxicity in Asian population is limited.

For this cohort, we plan to look at these topics:

1. proximal tubular dysfunction between TDF and non-TDF user
2. incidence and predictor of TDF related renal toxicity
3. TDF plasma concentrations
4. Pharmacokinetic of TDF when used with boosted DRV, boosted ATV, and boosted LPV in Thai population
5. Bone density and vitamin D in patients with and without hypophosphatemia.
6. Pharmacogenomic of TDF in Thai population

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old.
2. HIV RNA < 50 copies/ml (For ART-experienced group only).

Exclusion Criteria:

1. a history of Tc-99m DTPA allergy,
2. malnutrition (BMI <18m2),
3. amputation,
4. bed-ridden,
5. currently taking cotrimoxazole or cimetidine,
6. acute deterioration of renal function within the last 3 months,
7. serum creatinine > 1.5 mg/dl, or
8. pregnant/lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-NAT 006 participants (TDF +non TDF)and ARV naive population
  For TDF group, on TDF > 3 months HIV/HBV co-infected patients from COLD (Liver disease and HIV/HBV coinfection in the era of HAART) and TDF surveillance study
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
to validate eGFR Thai equation in HIV-infected adults | Blood specimens were drawn to assess plasma radioactivity at 5, 10, 20, 30, 60, 90, 120, 180, and 240 minutes post 99mTc-DTPA injection
  Test of diagnostic accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Praphan Phanuphak, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok, Thailand; Kearkiat Praditpornsilpa, MD, Principal Investigator — Renal division, Faculty of Medicine, Chulalongkorn University
Locations (1):
- HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok, Thailand

REFERENCES:
- [Result] Praditpornsilpa K, Avihingsanon A, Chaiwatanarat T, Chaiyahong P, Wongsabut J, Ubolyam S, Chulakadabba A, Avihingsanon Y, Ruxrungtham K, Tunsanga K, Eiam-Ong S, Phanuphak P. Comparisons between validated estimated glomerular filtration rate equations and isotopic glomerular filtration rate in HIV patients. AIDS. 2012 Sep 10;26(14):1781-8. doi: 10.1097/QAD.0b013e328356480d. PMID 22713478
- [Derived] Avihingsanon A, Kerr SJ, Ramautarsing RA, Praditpornsilpa K, Sophonphan J, Ubolyam S, Avihingsanon Y, Khovidhunkit W, Hiransuthikul N, Ruxrungtham K. The Association of Gender, Age, Efavirenz Use, and Hypovitaminosis D Among HIV-Infected Adults Living in the Tropics. AIDS Res Hum Retroviruses. 2016 Apr;32(4):317-24. doi: 10.1089/AID.2015.0069. Epub 2015 Oct 15. PMID 26413903
- [Derived] Punyawudho B, Thammajaruk N, Thongpeang P, Matthews G, Lewin SR, Burger D, Ruxrungtham K, Avihingsanon A. Population pharmacokinetics of tenofovir in HIV/HBV co-infected patients. Int J Clin Pharmacol Ther. 2015 Nov;53(11):947-54. doi: 10.5414/CP202386. PMID 26308175
- [Derived] Rungtivasuwan K, Avihingsanon A, Thammajaruk N, Mitruk S, Burger DM, Ruxrungtham K, Punyawudho B, Pengsuparp T. Influence of ABCC2 and ABCC4 polymorphisms on tenofovir plasma concentrations in Thai HIV-infected patients. Antimicrob Agents Chemother. 2015;59(6):3240-5. doi: 10.1128/AAC.04930-14. Epub 2015 Mar 23. PMID 25801567
- [Derived] Avihingsanon A, Jitmitraparp S, Tangkijvanich P, Ramautarsing RA, Apornpong T, Jirajariyavej S, Putcharoen O, Treeprasertsuk S, Akkarathamrongsin S, Poovorawan Y, Matthews GV, Lange JM, Ruxrungtham K; HIV-NAT125 study team. Advanced liver fibrosis by transient elastography, fibrosis 4, and alanine aminotransferase/platelet ratio index among Asian hepatitis C with and without human immunodeficiency virus infection: role of vitamin D levels. J Gastroenterol Hepatol. 2014 Sep;29(9):1706-14. doi: 10.1111/jgh.12613. PMID 24730732
- [Derived] Avihingsanon A, Apornpong T, Ramautarsing RA, Ubolyam S, Tangkijvanich P, Ananworanich J, Lange JM, Matthews G, Lewin SR, Ruxrungtham K; HIV-NAT 105 study team. Decline in serum 25 hydroxyvitamin D levels in HIV-HBV-coinfected patients after long-term antiretroviral therapy. Antivir Ther. 2014;19(1):41-9. doi: 10.3851/IMP2673. Epub 2013 Aug 23. PMID 23970149
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org